CLINICAL TRIAL: NCT03524456
Title: Home Blood Pressure Telemonitoring With an Adapted Device With SMS Capability in the Primary Care Setting
Brief Title: Home Blood Pressure SMS Telemonitoring in the Primary Care Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Peruana Cayetano Heredia (Other)
Responsible Party: Principal Investigator, Renzo Calderon, Researcher, Universidad Peruana Cayetano Heredia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 101180
Record Dates: First submitted 2018-05-02; First posted 2018-05-14 (Actual); Last update posted 2019-05-07 (Actual); Status verified 2019-05

CONDITIONS: Hypertension
Keywords: home blood pressure monitoring; sms; primary care
MeSH Terms: conditions — Hypertension; Smith-Magenis Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Home blood pressure monitoring (Experimental)
  Interventions: Other: Home blood pressure monitoring
- Usual monitoring (No Intervention)

INTERVENTIONS:
Other: Home blood pressure monitoring — Participants would use a blood pressure device at home, that sends the readings automatically to the health center via SMS. The physicians would use this tool for medication management or rescheduling visits.
  Arms: Home blood pressure monitoring

SUMMARY:
Hypertension is a public health problem worldwide, being responsible for 9.4 million deaths worldwide each year, as well as contributing to the burden of coronary, cerebrovascular, renal diseases, among others. The monitoring of blood pressure at home has gained importance in recent years, being related to adherence to treatment, as well as in the prevention of complications and optimization of pressure levels; In the same way, the use of information and communication technologies (ICT) in health has contributed to the improvement of communication systems by providing alternative tele-monitoring in this type of diseases.

Objective:

To evaluate the impact of tele-monitoring at home through tensiometers with integrated SMS system (text message), for the sending and recording of blood pressure and heart rate data in the primary care setting.

Methods:

A randomized controlled trial will be conducted, evaluating the intervention with the integrated blood pressure device with SMS capability, comparing it with the standard care. After a follow-up of 1 month, the effect on the values of systolic and diastolic blood pressure will be evaluated, as well as the adherence to treatment and complications related to arterial hypertension. A sample number of 20 participants per group was calculated, with a significance of 95% and a power of 80%, to detect a minimum significant difference of 10 mmHg.

DETAILED DESCRIPTION:
Objectives

Main Objective:

To evaluate the impact of the home blood pressure telemonitoring through a device with integrated SMS system, in blood pressure values in uncontrolled hypertensive patients.

Secondary objectives:

1. Compare adherence to treatment at the beginning and end of the follow-up between the group that uses integrated tele-monitoring with SMS and the usual monitoring.
2. Describe the experiences of the participants of the intervention group with the tele-monitoring system.

Methods

Study design: A randomized controlled trial will be conducted, which will be followed for 1 month. The main measurement will be to evaluate the difference in blood pressure levels in both groups at the end of the follow-up, the intervention group would use the device for 2 weeks.

Intervention group: Tele-monitoring with sphygmomanometer with SMS capacity Control group: Regular monitoring Follow-up time: 1 month Primary Outcome: Difference in systolic and diastolic blood pressure

Population: Hypertensive patients who attend a Primary Care Centers:

Condevilla Health Center

Inclusion criteria:

Older than 18 years-old. Diagnosis of hypertension more than 3 months ago. Not Controlled In antihypertensive medication

Exclusion criteria:

Patient with chronic kidney disease on hemodialysis or peritoneal dialysis. Pregnant women. Travel or change of address in the next 1 month.

Sample:

A sample of 20 participants per group was calculated, with a significance of 95% and a power of 80%, to show a difference of 10 mmHg, with a standard deviation of 10 and 12 according to the literature evaluated.

Assignment of groups:

A selection of patients will be made in the clinic of the health centers. If the inclusion and exclusion criteria are met, they will be invited to participate in the study, after accepting and signing the informed consent, a randomization will be made for complete blocks of 4 (2 controls, 2 interventions) until the total of 40 participants is reached, 20 in the intervention group and 20 in the control group.

Intervention group:

Participants will receive general education on hypertension and general care as well as training for the use of the tensiometer and a graphic guide provided by the manufacturer of the tensiometer.

The participants of the intervention group will receive a commercial blood pressure monitor "Omron Series 10®" which was integrated into an SMS messaging system using open hardware developing boards.

The measurement scheme will be programmed 4 times a day: 2 in the morning, and 2 in the evening with a 3-minute interval. If no record is received in 24hrs, specific reminder text messages will be sent to the patient, caregiver and/or relative, if after 2 days, there is no measurement, the patient will be contacted by phone and / or caregiver / family.

The SMS of the tensiometer to the information center will include the following data:

Systolic blood pressure Diastolic blood pressure Heart Rate Date Hour

The sphygmomanometer SMS will be sent to the information and monitoring center that will be hosted on a server in the cloud. The information and monitoring system will store blood pressure records and would be accessible to the primary care centers physicians, they would be free to any decision making regarding treatment adjustment or scheduling visits to the patients.

Development of tensiometer with SMS capacity:

An information acquisition and SMS sending station capable of capturing the tensiometer measurement will be developed using Arduino ® development cards.

The tensiometer will be linked through its USB interface to the development board, which in turn will send the blood pressure data automatically.

It should be mentioned that the operation of the tensiometer has not been altered, and remains the same as that recommended by the manufacturer. At the end of the pressure collection, the data will be sent automatically.

Control group:

The control group will receive the same educational session, and the usual monitoring in Health Centers will continue.

Outcome:

The difference in blood pressure values will be made, after 1 month of follow-up, under the same conditions as the initial measurement, as well as adherence to treatment, complications, and compliance with scheduled appointments during follow-up.

Analysis plan:

The primary statistical analysis will be a Mann-Whitney test of two independent samples comparing the change in blood pressure measured between the baseline and after 1 month of follow-up.

A secondary analysis of medication differences, adherence to treatment, complications, and fulfillment of appointments will be made, between the 2 study groups The level of significance will be given by a value of p <0.05.

Ethical aspects

Written informed consent will be requested from participants and caregivers / relatives.

The equipment will include a SIM card that will be recharged by the researchers of the study, as well as the cost of the equipment and the messaging packages will be covered by the researchers throughout the follow-up.

The present protocol will be presented to the CIE of the UPCH as well as to the CIE of the HNCH for its approval.

The data obtained will be confidential, the personal identifiers will be separated from the analysis database, which will be stored in a separate database, stored with a password to which only the researchers will have access. The SMS data will be sent in an encrypted way so that it can only be read by the information center.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years-old.
* Diagnosis of hypertension more than 3 months ago.
* Not Controlled hypertension
* In antihypertensive medication

Exclusion Criteria:

* Patient with chronic kidney disease on hemodialysis or peritoneal dialysis.
* Pregnant women.
* Travel or change of address in the next 4 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-04-09 (Actual); Primary Completion 2018-08-29 (Actual); Study Completion 2018-09-29 (Actual)

PRIMARY OUTCOMES:
Comparison of blood pressure diference before and after the intervention period between the control and intervention arm | 1 month
  Changes in the blood pressure levels would be compare in both study groups

CONTACTS AND LOCATIONS:
Locations (1):
- Centro de Salud Condevilla, Lima, Peru

IPD SHARING:
Plan to Share IPD: Undecided